CLINICAL TRIAL: NCT03391518
Title: Evaluation of Blood Flow Regulation With Laser Speckle Flowgraphy in Patients With Normal Tension Glaucoma and Healthy Individuals.
Brief Title: Evaluation of Blood Flow Regulation With Laser Speckle Flowgraphy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Augenabteilung Allgemeines Krankenhaus Linz (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LSFG_WDT
Record Dates: First submitted 2017-12-30; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Low Tension Glaucoma
MeSH Terms: conditions — Low Tension Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Water drinking test — Ingestion of 800 ml water in less than 5 minutes.

SUMMARY:
The study includes Caucasian patients with diagnosis of normal tension glaucoma and age- and sex-matched healthy individuals. Measurements of optic nerve head blood flow will be performed with laser speckle flowgraphy (LSFG). Also, the intraocular pressure (IOP), systolic and diastolic blood pressure, heart rate (HR), mean arterial pressure (MAP) as well as ocular perfusion pressure (OPP) will be evaluated. After baseline measurements individuals will be asked to ingest 800 ml of water in less than five minutes. Measurements will be repeated after 15, 30 and 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* presence of glaucomatous optic disc changes in biomicroscopy and visual field defects or abnormal circumpapillary retinal nerve fibre layer (RNFL) thinning (evaluated by OCT as defined by the on-board software)
* IOP ≤ 21mmHg without therapy
* normal open angle in a gonioscopic examination
* age > 40 years

Exclusion Criteria:

* IOP > 21 mmHg in patients' history
* ametropia > 6 diopters
* cataract with severity greater than grade 2 of the lens opacities classification system (LOCS) classification
* presence of corneal opacities
* uncontrolled hypertension with systolic blood pressure (SBP) > 165mmHg and/or diastolic blood pressure (DBP) > 100mmHg

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2018-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in ONH blood flow induced by water drinking test | baseline, after 15, 30 and 45 minutes
  ONH blood flow evaluated by laser speckle flowgraphy

CONTACTS AND LOCATIONS:
Locations (1):
- AKh Linz, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No